CLINICAL TRIAL: NCT03355287
Title: Assessing the Impact of Soil Iron Intake From Teff Flour on Iron Status in Infants in Ethiopia.
Brief Title: Iron Status in Infants in Ethiopia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Addis Ababa University (Other); HarvestPlus (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Dr.Prof., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Eth_Teff_Iron
Record Dates: First submitted 2017-11-13; First posted 2017-11-28 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Aluminium Intoxication
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditionally Threshed Teff (TTT) (Placebo Comparator): The control group will consume injera based on teff threshed under the hooves of cattle. We plan to have a certain number of teff flour suppliers, where the teff is traditionally threshed and contains at least 50 mg Fe per 100 g flour.
  Interventions: Other: Traditionally Threshed Teff (TTT)
- Lab Threshed Teff (LTT) (Experimental): The intervention group will consume injera based on teff flour that has been lab threshed using a modern teff threshing machine.
  Interventions: Other: Lab Threshed Teff (LTT)
- Fortified Lab Threshed Teff (FTT) (Active Comparator): This arm will be the positive control group consuming Ferrous Sulphate drops ( with injera that consist of lab-threshed teff. The Fe drops have to be consumed with the meal and will provide an additional 6 mg of Ferrous sulfate to the diet of the children.
  Interventions: Other: Fortified Lab Threshed Teff (FTT)

INTERVENTIONS:
Other: Traditionally Threshed Teff (TTT) — The intervention will take place for 7 months in Debre Zeit where the the arm will be fed injera based on teff that are threshed traditionally
  Arms: Traditionally Threshed Teff (TTT)
Other: Lab Threshed Teff (LTT) — The intervention will take place for 7 months in Debre Zeit where this arm will be fed injera from teff that is threshed using a modern thresher.
  Arms: Lab Threshed Teff (LTT)
Other: Fortified Lab Threshed Teff (FTT) — The intervention will take place for 7 months in Debre Zeit where this arm will be fed injera from teff that is threshed using a modern thresher. In addition, they will receive Ferrous sulfate drops
  Arms: Fortified Lab Threshed Teff (FTT)

SUMMARY:
To assess the impact of soil iron intake from teff flour on iron status in infants in Debre Zeit, Ethiopia.

DETAILED DESCRIPTION:
Rationale: Teff (Eragrostis Teff), a major staple crop in several areas of Ethiopia, is of special relevance to Fe biofortifcation as it provides the population with a regular high consumption of contaminant soil Fe due to the traditional threshing procedure under the hooves of the cattle. The bioavailability of soil Fe, and hence its contribution to Fe requirements, is unknown. Data on the bioavailability of soil Fe would clarify to what extent the soil Fe can be considered as a source of absorbable Fe. This information is important in order to establish dietary advice and is essential for the development of iron biofortification (and fortification) policies related to Fe nutrition in Ethiopia.

Objective: The overall objective of the project is to generate data to target and tailor biofortification approaches in Ethiopia by an intervention trial assessing the impact of soil Fe intake from teff consumption on Fe status.

Study design: The intervention trial will be a 7 months partially blinded, randomized control trial (RCT) with the following three arms: control-group consuming injera based on traditionally threshed teff (average Fe content 50 mg/100g flour), 2) intervention group consuming injera based on lab-threshed teff (average Fe content 6.65 mg/100g flour), 3) positive control group consuming the lab-threshed teff together with ferrous sulphate iron drops (additional Fe from the drops = 6 mg).

Study population: 315 children between 18-36 months of age living in Debre Zeit and surrounding areas will be enrolled.

Main study parameters/endpoints: The impact of soil Fe in teff on Fe status will be assessed by measuring the Fe status, prevalence of Fe deficiency and Fe deficiency anemia at baseline, midpoint and endpoint. To assess Fe status, Hemoglobin (Hb), Plasma Ferritin (PF), Soluble Transferrin Receptor (sTfR), C- Reactive Protein(CRP) and Alpha 1B glycoprotein (AGP) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* 18-36 months of age (at screening)
* The child is able to eat at least two injera meals per day
* The informed consent form has been read and signed by the caregiver (or has been read out to the caregiver in case of illiteracy)

Exclusion Criteria:

* Severely deficient in Hb (<70g/L)
* Severe underweight (weight for age Z score < -3),
* Severe wasting (weight for height Z score < -3)
* Chronic or acute illness or other conditions that in the opinion of the Principle Investigator (PI) or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participants taking part in other studies requiring the drawing of blood
* Not planning long-term residence in study site

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 315 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Change in Haemoglobin | Three collection points - First collection point at screening, second collection point at mid point (3.5 months after start of intervention) and third collection point at the end point ( end of the 7 months of the intervention)
  Iron status
Change in Ferritin | Two collection points - First collection point at screening, second collection point at the end of the study ( 7 months after the intervention start )
  Iron status
Change in Soluble Transferrin Receptor (sTfR) | Two collection points - First collection point at screening, second collection point at the end of the study ( 7 months after the intervention start )
  Iron status
Change in C-Reactive Protein (CRP) | Two collection points - First collection point at screening, second collection point at the end of the study ( 7 months after the intervention start )
  Inflammation
Change in Alpha 1-Acid Glycoprotein (AGP) | Two collection points - First collection point at screening, second collection point at the end of the study ( 7 months after the intervention start )
  Inflammation

SECONDARY OUTCOMES:
Change in Aluminium (Al) levels | Two collection points - First collection point at screening, second collection point at the end of the study ( 7 months after the intervention start )
  Measuring Al in plasma
Change in Aluminium (Al) levels | Three collection points - First collection point at the first day of the study, Second collection point during mid point ( 3.5 months after start of the intervention, and third collection point at the end of the intervention ( end of 7th month)
  Measuring Al in hair and nail
Change in Anthropometric measurements | Three collection points - First collection point during screening, Second collection point during mid point ( 3.5 months after start of the intervention, and third collection point at the end of the intervention ( end of 7th month)
  Weight in kg
Change in Anthropometric measurements | Three collection points - First collection point during screening, Second collection point during mid point ( 3.5 months after start of the intervention, and third collection point at the end of the intervention ( end of 7th month)
  Height in cm
Teff flour | Through study completion, an average of 7 months
  Iron concentration
Teff flour | Through study completion, an average of 7 months
  Phytate content
Morbidity | Through study completion, an average of 7 months
  Any sickness arising due to the consumption of the meals
Injera consumption | Through study completion, an average of 7 months
  Amount of injera consumed by the child in each meal
2 day weighted food record | Through study completion, an average of 7 months
  To estimate the amount of different foods consumed by the child

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Dr. PhD, Principal Investigator — Swiss Federal Institute of Technology, ETH Zurich, Switzerland; Kaleab Baye, PhD, Principal Investigator — Assistant Professor and Head, Center for Food Science and Nutrition, Addis Ababa Univeristy, Ethiopia
Locations (2):
- Center for Food Science and Nutrition, Addis Ababa University, Addis Ababa, Ethiopia
- Swiss Federal Institute of Technology ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No